CLINICAL TRIAL: NCT04580849
Title: Telerehabilitation Using a Dance Intervention in People With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Principal Investigator, Aline de Souza Pagnussat, Principal Investigator, Federal University of Health Science of Porto Alegre
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TELEDANCE
Record Dates: First submitted 2020-10-01; First posted 2020-10-09 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Telerehabilitation

STUDY DESIGN:
Intervention Model Description: individuals with parkinson's disease and healthy control individuals will be assigned to the same online dance class via zoom platform.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- telerehabilitation with dance (Parkinson's) (Experimental): This group will receive dance classes online during 60 minutes, twice a week for 8 weeks.
  Interventions: Other: telerehabilitation with dance
- telerehabilitation with dance (Healthy controls) (Active Comparator): This group will receive dance classes online during 60 minutes, twice a week for 8 weeks.
  Interventions: Other: telerehabilitation with dance

INTERVENTIONS:
Other: telerehabilitation with dance — Dance classes will be provided through a online platform. Each class will last 60 minutes, twice a week, during 8 weeks.

SUMMARY:
The aim of this study is to verify the feasibility of a telerehabilitation approach with dance in people with parkinson's disease.

DETAILED DESCRIPTION:
This is a feasibility study that aims to investigate the safety and efficacy of dance classes via an online platform in people with and without Parkinson's Disease. The intervention will last 2 months and the classes will be conducted twice a week (60 minutes) using the Zoom platform. Evaluations will be performed before and after the intervention by means of the Zoom platform as well and will include questionnaires of quality of life, depression, anxiety, and activities of daily living.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with and without parkinson's disease according London Brain Bank Criteria
* Minimal cognitive ability to understand commands (MMSE)
* Able to stand at least 10 minutes with or without support
* Dopamine medication stable at least 6 weeks before the beginning of the study
* Portable device and internet connection

Exclusion Criteria:

* Severe visual or auditive disturbances
* Neurological disease (other than parkinson's for those included) or severe neuromuscular disorders that prejudice the proposed activities

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-09-05 (Actual); Primary Completion 2020-10-05 (Actual); Study Completion 2020-12-05 (Actual)

PRIMARY OUTCOMES:
feasibility (adherence rates) | 10 weeks
  To assess the feasibility of the study design and procedures. The adherence rate will be calculated by the total number of patients who completed the full course of intervention divided by the total number of patients included at the beginning.

SECONDARY OUTCOMES:
feasibility (patients opinions) | 10 weeks
  Semi structured interviews will involve gaining patients opinions on the strengths and weaknesses of the intervention
feasibility (safety and usability) | 10 weeks
  The researches will follow all patients during the intervention regarding safety (i.e. falls) and usability (i.e. internet connection)
Parkinson's Disease Questionnaire-8 (PDQ-8) | Change from Pre to Post treatment (10 weeks)
  The PDQ-8 is a short-form version to assess quality of life in persons with Parkinson's disease. Each question is scored from 0-4 points and the scores are summed and given as a percentage score (0-100). The higher the score, the worse the patient's condition.
36-Item Short Form Survey (SF-36) | Change from Pre to Post treatment (10 weeks)
  The SF-36 measures health-related quality of life. This questionnaire has 36-item measure divided into 8 subscales - each subscale can be used independently. Each of the 8 summed scores is transformed into a scale from 0 (negative health) to 100 (positive health)
Hospital Anxiety and Depression Scale (HADS) | Change from Pre to Post treatment (10 weeks)
  The scale is used to identify depression and anxiety and presents 14 items. The total score is out of 42. The higher scores indicate greater levels of anxiety and depression.
Unified Parkinson's Disease Rating Scale (UPDRS) Part I | Change from Pre to Post treatment (10 weeks)
  The Part I concerns about non-motor experiences of daily living (e.g. anxiety and depression). This scale has 13 questions and all items have 5 response options. Higher scores indicate greater impact of PD symptoms.
Activities-Specific Balance (ABC) Scale | Change from Pre to Post treatment (10 weeks)
  Self-reported questionnaire measuring self-efficacy in performing activities without losing balance. The ABC Scale consists of 16 questions that require the patient to rate their confidence on a scale from 0% to 100%. The higher the percentage, the higher level of physical functioning.
Five Times Sit to Stand Test (FTSTS) | Change from Pre to Post treatment (10 weeks)
  The test assess the functional mobility strength of lower extremity (measured by the time to complete the test). The higher the time to complete the test, the lower the performance.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal de Ciências da Saúde de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No